CLINICAL TRIAL: NCT01687725
Title: Renal Denervation in Treatment Resistant Hypertension
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: RD-TRH
Record Dates: First submitted 2012-09-13; First posted 2012-09-19 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal denervation: Renal denervation using Symplicity Catheter system
  Interventions: Device: Renal denervation using Symplicity Catheter system

INTERVENTIONS:
Device: Renal denervation using Symplicity Catheter system — percutaneous selective renal sympathetic nerve ablation with the use of the Symplicity Catheter system

SUMMARY:
In patients with treatment resistant hypertension renal nerve ablation emerged as an effective interventional approach of treating hypertensive disease with a progressively increasing fall in blood pressure. Decreased activity of the sympathetic nervous system is one of the major underlying pathogenetic mechanism of the fall in blood pressure but the precise mechanisms that causes the fall in blood pressure in the short-term and, in particular, long-term remains elusive. The objective of the study is to understand the pathogenetic mechanisms of renal denervation beyond the reduced activity of the sympathetic nervous system. In 100 hypertensive patients most advanced technology will be applied, before and repeatedly after renal denervation, throughout the follow-up period of 1 year. Systemic activity of the renin angiotensin aldosterone system, renal perfusion (by MRI spin labeling technique), local activity of the renin angiotensin system in the kidney (urinary angiotensinogen concentrations), sodium excretion and total sodium content (23 Na-MRI technique) and vascular remodelling of small (retinal arterioles 50 - 150 µm) and large arteries (carotid - femoral pulse wave velocity and augmentation index, both measured over 24 hours) will be assessed. Identification of the pathogenetic mechanisms involved in the fall in blood pressure after renal denervation may help to identify those hypertensive patients that profit most from renal nerve ablation in terms of blood pressure reduction.

The investigators propose the following hypotheses why a progressive decrease in blood pressure happens, in addition to the decreased activity of the central nervous system, after renal nerve ablation:

Short term effects:

A)Preservation of renal function and perfusion B)Reduction of local RAS activity in the kidney C)Exaggerated sodium excretion immediately after renal nerve ablation

Long term effects:

D)Decrease of total sodium content after 6 and 12 months E)Improvement of vascular wall properties after 6 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* treatment resistant hypertension
* male of female aged over 18 years
* written informed consent
* agreement to attend all study visits as planned in the protocol

Exclusion Criteria:

* chronic kidney disease 3 - 5
* any contradictions for MRI
* claustrophobia
* strabismus
* severe ocular diseases
* history of epilepsia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: treatment resistant hypertensive adults
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
office BP | baseline, 6 months
  change in office blood pressure from baseline to 6 months post-renal denervation
24-ABPM | baseline, 6 months
  change in 24 hour ambulatory blood pressure (ABPM) from baseline to 6 months post-renal denervation
Magnetic resonance imaging (MRI) | baseline, 3 and 6 months
  * change in total sodium content measured by MRI from baseline to 6 months post-renal denervation
  * change in renal perfusion measured by MRI from baseline to 3 months post-renal denervation
Albuminuria | baseline, 6 months
  change in urinary albumin/creatinine ratio from baseline to 6 months post-renal denervation
Systemic RAS activity | baseline, 6 months
  * change in sodium, potassium and creatinine from baseline to 6 months post-renal denervation
  * change in aldosterone excretion from baseline to 6 months post-renal denervation
  * change in sodium/potassium ratio from baseline to 6 months post-renal denervation
  * change in plasma renin activity and angiotensin II concentration at least 30 minutes of rest in a supine position and immediately after standing from baseline to 6 months post-renal denervation
Vascular structure and function of large and small arteries | baseline, 6 months
  * change in flow-mediated vasodilation (FMD)from baseline to 6 months post-renal denervation
  * change in scanning laser Doppler flowmetry (SLDF) from baseline to 6 months post-renal denervation
  * change in funduscopy from baseline to 6 months post-renal denervation
  * change in pulse wave analysis (PWA) from baseline to 6 months post-renal denervation
  * change in pulse wave velocity (PWV) from baseline to 6 months post-renal denervation
  * change in urinary albumine/creatinine ratio (UACR) of the morning spot urine sample from baseline to 6 months post-renal denervation
Local RAS activity | baseline, 6 months
  change in urinary angiotensinogen concentration from the morning spot urine from baseline to 6 months post-renal denervation

SECONDARY OUTCOMES:
BP | 3 and 12 months
  * change in office BP from baseline to 3 and 12 months post-renal denervation
  * change in 24 hour ABPM from baseline to 3 and 12 months post-renal denervation
MRI | 1 day and 12 months
  * change in total sodium content measured by MRI from baseline to 12 months post-renal denervation
  * change in renal perfusion measured by MRI spin labelling technique from baseline to 1 day post-renal denervation
Local RAS activity | 1 day, 3 and 12 months
  change urinary angiotensinogen concentration from the morning spot urine from baseline to 1 day, 3 and 12 months post-renal denervation
Systemic RAS activity | 1 day, 3 and 12 months
  * change in sodium potassium and creatinine from baseline to 1 day, 3 and 12 months post-renal denervation
  * change in aldosterone excretion from baseline to 1 day, 3 and 12 months post-renal denervation
  * change in sodium/potassium ratio from baseline to 1 day, 3 and 12 months post-renal denervation
  * change in plasma renin activity and angiotensin II concentration at least 30 minutes of rest in a supine position and immediately after standing from baseline to 1 day, 3 and 12 months post-renal denervation
Albuminuria | 3 and 12 months
  - change in albuminuria from baseline to 3 and 12 months post-renal denervation
Vascular structure and function of large and small arteries | 3 and 12 months
  * change in flow mediated vasodilation (FMD) from baseline to 12 months post-renal denervation
  * change in scanning laser Doppler flowmetry (SLDF) from baseline to 12 months post-renal denervation
  * change in funduscopy from baseline to 3 and 12 months post-renal denervation
  * change in pulse wave analysis (PWA) from baseline to 12 months post-renal denervation
  * change in pulse wave velocity (PWV) from baseline to 12 months post-renal denervation
  * change in urinary albumine/creatinine ratio of the morning spot urine sample from baseline to 3 and 12 months post-renal denervation

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, Principal Investigator — University of Erlangen-Nürnberg
Locations (2):
- Germany (2):
  - Clinical Research Unit, Department of Nephrology and Hypertension, University of Erlangen-Nürnberg, Erlangen
  - Klinik für Innere Medizin, Kardiologie, Angiologie und Internistische Intensivmedizin, Universitätsklinikum des Saarlandes, Homburg/Saar

REFERENCES:
- [Background] Ott C, Harazny JM, Schmid A, Ditting T, Veelken R, Bladowski M, Michelson G, Uder M, Schmieder RE. Retinal microperfusion after renal denervation in treatment-resistant hypertensive patients. Clin Res Cardiol. 2015 Sep;104(9):782-9. doi: 10.1007/s00392-015-0845-0. Epub 2015 Apr 28. PMID 25916737
- [Background] Ott C, Mahfoud F, Schmid A, Ewen S, Toennes SW, Meyer MR, Helfer AG, Maurer HH, Ditting T, Veelken R, Zivanovic I, Uder M, Bohm M, Schmieder RE. The effect of renal denervation in moderate treatment-resistant hypertension with confirmed medication adherence. J Hypertens. 2016 Dec;34(12):2475-2479. doi: 10.1097/HJH.0000000000001110. PMID 27607458
- [Background] Ott C, Mahfoud F, Schmid A, Toennes SW, Ewen S, Ditting T, Veelken R, Ukena C, Uder M, Bohm M, Schmieder RE. Renal denervation preserves renal function in patients with chronic kidney disease and resistant hypertension. J Hypertens. 2015 Jun;33(6):1261-6. doi: 10.1097/HJH.0000000000000556. PMID 25923731
- [Derived] Guenes-Altan M, Schmid A, Kannenkeril D, Linz P, Ott C, Bosch A, Schiffer M, Uder M, Schmieder RE. Skin sodium content as a predictor of blood pressure response to renal denervation. Hypertens Res. 2024 Feb;47(2):361-371. doi: 10.1038/s41440-023-01450-4. Epub 2023 Oct 25. PMID 37880499
- [Derived] Bosch A, Schmid A, Ott C, Kannenkeril D, Karg MV, Ditting T, Veelken R, Uder M, Schmieder RE. Copeptin Levels in Patients With Treatment-Resistant Hypertension Before and 6 Months After Renal Denervation. Am J Hypertens. 2020 Feb 22;33(2):182-189. doi: 10.1093/ajh/hpz155. PMID 31555795
- [Derived] Ott C, Kopp C, Dahlmann A, Schmid A, Linz P, Cavallaro A, Hammon M, Ditting T, Veelken R, Uder M, Titze J, Schmieder RE. Impact of renal denervation on tissue Na+ content in treatment-resistant hypertension. Clin Res Cardiol. 2018 Jan;107(1):42-48. doi: 10.1007/s00392-017-1156-4. Epub 2017 Aug 28. PMID 28845508
- [Derived] Schmieder RE, Ott C, Schmid A, Friedrich S, Kistner I, Ditting T, Veelken R, Uder M, Toennes SW. Adherence to Antihypertensive Medication in Treatment-Resistant Hypertension Undergoing Renal Denervation. J Am Heart Assoc. 2016 Feb 12;5(2):e002343. doi: 10.1161/JAHA.115.002343. PMID 26873693
- [Derived] Ott C, Schmid A, Toennes SW, Ditting T, Veelken R, Uder M, Schmieder RE. Central pulse pressure predicts BP reduction after renal denervation in patients with treatment-resistant hypertension. EuroIntervention. 2015 May;11(1):110-6. doi: 10.4244/EIJV11I1A19. PMID 25982653
- [Derived] Ott C, Mahfoud F, Schmid A, Ditting T, Veelken R, Ewen S, Ukena C, Uder M, Bohm M, Schmieder RE. Improvement of albuminuria after renal denervation. Int J Cardiol. 2014 May 1;173(2):311-5. doi: 10.1016/j.ijcard.2014.03.017. Epub 2014 Mar 15. PMID 24681017
- [Derived] Ott C, Mahfoud F, Schmid A, Ditting T, Sobotka PA, Veelken R, Spies A, Ukena C, Laufs U, Uder M, Bohm M, Schmieder RE. Renal denervation in moderate treatment-resistant hypertension. J Am Coll Cardiol. 2013 Nov 12;62(20):1880-6. doi: 10.1016/j.jacc.2013.06.023. Epub 2013 Jul 10. PMID 23850901